CLINICAL TRIAL: NCT01964976
Title: Nesina Tablets Special Drug Use Surveillance Type 2 Diabetes Mellitus: Combination Therapy With Biguanides
Brief Title: Alogliptin Tablets Special Drug Use Surveillance Type 2 Diabetes Mellitus: Combination Therapy With Biguanides
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 121-014; JapicCTI-132282 (Registry Identifier: JapicCTI); JapicCTI-R150790 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-02

CONDITIONS: Surveillance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Alogliptin + Biguanides: All participants who received alogliptin 25 milligram (mg), tablets, orally, once daily for up to 12 months along with biguanide or without biguanide within 3 months from the start of administration of alogliptin and during the treatment period of alogliptin as per routine clinical practice were observed in this study.

SUMMARY:
To examine the safety and efficacy of long-term combination therapy with alogliptin (Nesina) and biguanides in participants with type 2 diabetes mellitus who responded inadequately to treatment with biguanides in addition to diet therapy and exercise therapy.

DETAILED DESCRIPTION:
This is a special drug use surveillance on long-term use of alogliptin with a 1-year (12-month) observational period, designed to investigate the safety and efficacy of long-term combination therapy with alogliptin and biguanides in participants with type 2 diabetes mellitus in the routine clinical setting.

Participants diagnosed with type 2 diabetes mellitus who responded inadequately to treatment with biguanides in addition to diet therapy and exercise therapy will be enrolled. The planned sample size is 1,000.

The usual adult dosage for oral use is 1 alogliptin tablet (25 mg) once daily.

ELIGIBILITY:
Inclusion Criteria:

* Participants who did not adequately respond to the following treatment • Treatment with biguanides in addition to diet therapy and exercise therapy

Exclusion Criteria:

* Participants contraindicated for Nesina

  1. Participants with severe ketosis, diabetic coma or precoma, or type 1 diabetes mellitus [these participants require prompt adjustment of hyperglycemia by fluid infusion and insulin, and hence use of Nesina is not appropriate].
  2. Participants with severe infection, pre- or post-operative patients, or patients with serious traumatic injury [blood glucose control by insulin injection is desirable for these participants, and hence use of Nesina is not appropriate].
  3. Participants with a history of hypersensitivity to any ingredient of Nesina.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with type 2 diabetes mellitus who have been examined at a medical institution
Sampling Method: Non-Probability Sample
Enrollment: 1096 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Postmarketing Group Manager, Study Chair — Takeda
Locations (1):
- Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 207 investigative sites in Japan from 01 July 2011 to 31 December 2014.
Pre-assignment Details: Participants with type 2 diabetes mellitus started treatment with alogliptin as per routine clinical practice were observed. As per protocol, participants were enrolled in 1 observational group at the start and were divided into 2 groups based on biguanide use for analysis of safety endpoints. Participant flow data was collected for overall arm.
Groups:
- All Population: All participants who received alogliptin 25 milligram (mg), tablets, orally, once daily for up to 12 months along with biguanide or without biguanide within 3 months from the start of administration of alogliptin and during the treatment period of alogliptin as per routine clinical practice were observed in this study.
Period: Overall Study
Arm/Group | All Population
Started | 1096 (Data reports overall population,since data not collected separately per arm as specified in protocol)
Completed | 1065
Not Completed | 31
Not completed — Protocol Violation | 31

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who completed the study and had safety data available.
Groups:
- Alogliptin + Biguanides: Alogliptin 25 milligram (mg), tablets, orally, once daily for up to 12 months in participants who received a biguanide within 3 months from the start of administration of alogliptin and during the treatment period of alogliptin as per routine clinical practice were observed in this study.
- Alogliptin + Other: Alogliptin 25 mg, tablets, orally, once daily for up to 12 months in participants who did not receive a biguanide within 3 months from the start of administration of alogliptin or during the treatment period of alogliptin as per routine clinical practice were observed in this study.
- Total: Total of all reporting groups
Arm/Group | Alogliptin + Biguanides | Alogliptin + Other | Total
Number analyzed (Participants) | 954 | 109 | 1063
Age, Customized [Number; unit: participants]
  Less than (<) 65 years | 539 | 68 | 607
  Greater than or equal to (>=) 65 years | 415 | 41 | 456
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 388 | 37 | 425
  Male | 566 | 72 | 638
Time from Diagnosis of Type 2 Diabetes [Number; unit: participants]
  <2 years | 114 | 16 | 130
  >=2 to <5 years | 169 | 20 | 189
  >=5 to <10 years | 218 | 19 | 237
  >=10 years | 254 | 27 | 281
  Unknown | 199 | 27 | 226
Body Mass Index [Number; unit: participants]
  <25 kilogram per square meter (kg/m^2) | 345 | 35 | 380
  >=25 kg/m^2 | 410 | 45 | 455
  Unknown | 199 | 29 | 228
Waist Circumference [Number; unit: participants]
  <85 centimeter (cm) (Male) | 25 | 5 | 30
  >=85 cm (Male) | 90 | 4 | 94
  Unknown (Male) | 451 | 63 | 514
  <90 cm (Female) | 37 | 4 | 41
  >=90 cm (Female) | 33 | 3 | 36
  Unknown (Female) | 318 | 30 | 348
Pregnancy Status [Number; unit: participants] — This baseline characteristic was analyzed only in female participants.
  participants
    Not pregnant | 388 | 37 | 425
    Pregnant | 0 | 0 | 0
Healthcare Category [Number; unit: participants] — Participants were categorized as outpatient, inpatient, and outpatient and inpatient (participants who were both outpatient and inpatient during some point at the time and 3 months prior to enrollment).
  participants
    Outpatient | 920 | 102 | 1022
    Inpatient | 2 | 1 | 3
    Outpatient and inpatient | 32 | 6 | 38
Degree of Renal Dysfunction [Number; unit: participants] — Estimated glomerular filtration rate (eGFR) was calculated using variables of gender, age at the start of treatment, and serum creatinine values, and severity was determined based on the following categories. If the serum creatinine value at the start of treatment was not listed, the severity was listed as "unknown." Normal: >=90 milliliter per minute (mL/min)/1.73^2, Mild: >=60 mL/min/1.73^2 to <90 mL/min/1.73^2 Moderate: >=30 mL/min/1.73^2 to <60 mL/min/1.73^2, Severe: <30 mL/min/1.73^2. eGFR = 194 * Cr^-1.094 * (age)^-0.287 (* 0.739 if female), where Cr is serum creatinine.
  participants
    Normal | 213 | 12 | 225
    Mild | 359 | 50 | 409
    Moderate | 135 | 13 | 148
    Severe | 3 | 0 | 3
    Unknown | 244 | 34 | 278
History of Allergy [Number; unit: participants]
  Had allergy | 773 | 84 | 857
  Did not have allergy | 92 | 10 | 102
  Unknown | 89 | 15 | 104
Health-related Complications [Number; unit: participants]
  Had complications | 862 | 91 | 953
  Had no complications | 92 | 18 | 110
Diabetic complications [Number; unit: participants]
  Had complications | 206 | 20 | 226
  Had No Complications | 748 | 89 | 837
Breakdown of diabetic complications [Number; unit: participants] — This baseline characteristic was analyzed only in participants who had diabetic complications. Participants may be represented in more than 1 category.
  participants
    Diabetic nephropathy | 110 | 12 | 122
    Diabetic retinopathy | 91 | 10 | 101
    Diabetic neuropathy | 83 | 8 | 91
Complications of Hypertension [Number; unit: participants]
  Had complications | 567 | 54 | 621
  Had no complications | 387 | 55 | 442
Complications of Dyslipidemia [Number; unit: participants]
  Had complications | 623 | 69 | 692
  Had no complications | 331 | 40 | 371
Complications of Hyperuricemia [Number; unit: participants]
  Had complications | 69 | 14 | 83
  Had no complications | 885 | 95 | 980
Complications of Liver Damage [Number; unit: participants]
  Had complications | 203 | 20 | 223
  Had no complications | 751 | 89 | 840
Breakdown of Complications of Liver Damage [Number; unit: participants] — Liver damage complications were categorized as hepatic steatosis, hepatitis alcoholic, chronic hepatitis, hepatic cirrhosis and any other complications related to liver damage. This baseline characteristic was analyzed only in participants who had complications of liver damage. Participants may be represented in more than 1 category.
  participants
    Hepatic steatosis | 158 | 15 | 173
    Hepatitis alcoholic | 23 | 5 | 28
    Chronic hepatitis | 15 | 5 | 20
    Hepatic cirrhosis | 2 | 1 | 3
    Other | 7 | 0 | 7
Degree of Hepatic Dysfunction [Number; unit: participants] — Severity was determined using aspartate aminotransferase (AST) or alanine transaminase (ALT) values at the start of treatment with alogliptin. For the assessment of severity, the following categories were used and a higher severity grade for either AST or ALT serum levels was adopted. Normal: <50 international units per liter (IU/L), Grade 1: >=50 to <100 IU/L, Grade 2: >=100 to <500 IU/L, and Grade 3: >=500 IU/L.
  participants
    Normal | 597 | 65 | 662
    Grade 1 | 81 | 13 | 94
    Grade 2 | 21 | 1 | 22
    Unknown | 255 | 30 | 285
Complications of Renal Damage [Number; unit: participants]
  Had complications | 114 | 12 | 126
  Had No Complications | 840 | 97 | 937
Breakdown of Complications of Renal Damage [Number; unit: participants] — Renal damage complications were categorized as nephrotic syndrome, glomerulonephritis, renal failure chronic and any other complications related to renal damage. This baseline characteristic was analyzed only in participants who had renal damage complications. Participants may be represented in more than 1 category.
  participants
    Nephrotic syndrome | 1 | 0 | 1
    Glomerulonephritis | 1 | 0 | 1
    Renal failure chronic | 2 | 0 | 2
    Other | 110 | 12 | 122
Complications of Heart Disease [Number; unit: participants]
  Had complications | 103 | 7 | 110
  Had no complications | 851 | 102 | 953
Breakdown of Complications of Heart Disease [Number; unit: participants] — Heart disease complications were categorized as cardiac failure, myocardial infarction, angina pectoris, and any other complications related to heart disease. This baseline characteristic was analyzed only in participants who had heart disease complications. Participants may be represented in more than 1 category.
  participants
    Cardiac failure | 19 | 1 | 20
    Myocardial infarction | 24 | 1 | 25
    Angina pectoris | 49 | 3 | 52
    Other | 24 | 2 | 26
Complications of Heart Failure [Number; unit: participants]
  Had complications | 19 | 1 | 20
  Had no complications | 935 | 108 | 1043
New York Heart Association (NYHA) Heart Failure Classification [Number; unit: participants] — NYHA functional classification ranges from Class I (participants with cardiac disease but without resulting limitations of physical activity), Class II (participants with cardiac disease resulting in slight limitation of physical activity), Class III (participants with cardiac disease resulting in marked limitation of physical activity), Class IV (participants with cardiac disease resulting in inability to carry on any physical activity without discomfort). This baseline measure was analyzed only for participants who had complications of heart failure.
  participants
    NYHA Class I | 13 | 0 | 13
    NYHA Class II | 5 | 0 | 5
    NYHA Class IV | 1 | 1 | 2
Complications of Stroke-related Disease [Number; unit: participants]
  Had complications | 58 | 5 | 63
  Had no complications | 896 | 104 | 1000
Breakdown of Complications of Stroke-related Disease [Number; unit: participants] — This baseline characteristic was analyzed only in participants who had complications of stroke-related disease.
  participants
    Cerebral infarction | 57 | 5 | 62
    Cerebral hemorrhage | 1 | 0 | 1
Complications of Allergic Disease [Number; unit: participants]
  Had complications | 66 | 7 | 73
  Had no complications | 888 | 102 | 990
Complications of Malignant Tumor [Number; unit: participants]
  Had complications | 18 | 6 | 24
  Had no complications | 936 | 103 | 1039
Other Complications [Number; unit: participants] — Participants who had complications other than diabetic, hypertension, dyslipidemia, hyperuricemia, liver damage, renal damage, heart disease, heart failure, stroke-related disease, allergic disease, and malignant tumor were analyzed in this measure.
  participants
    Had complications | 315 | 38 | 353
    Had no complications | 639 | 71 | 710
Presence of Medical History [Number; unit: participants]
  Had medical history | 150 | 30 | 180
  Did not have medical history | 694 | 68 | 762
  Unknown | 110 | 11 | 121
History of Alcohol Consumption [Number; unit: participants] — In this measure, participants responded whether they consumed alcohol-containing beverages nearly every day or not.
  participants
    Yes | 231 | 26 | 257
    No | 573 | 60 | 633
    Unknown | 150 | 23 | 173
Smoking Classification [Number; unit: participants]
  Never Smoked | 442 | 45 | 487
  Current Smoker | 167 | 18 | 185
  Ex-smoker | 162 | 15 | 177
  Unknown | 183 | 31 | 214
Glycosylated Hemoglobin (HbA1c) Level [Number; unit: participants]
  HbA1c <6.0 percent (%) | 12 | 5 | 17
  HbA1c >=6.0% to <7.0% | 177 | 16 | 193
  HbA1c >=7.0% to <8.0% | 381 | 43 | 424
  HbA1c >=8.0% | 341 | 35 | 376
  Unknown | 43 | 10 | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Adverse Drug Reactions
Description: Adverse drug reactions are defined as adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment. AEs are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug. The safety analysis was planned to be assessed in alogliptin + biguanides and alogliptin + other arm separately.
Time Frame: Baseline up to 12 months
Population: The safety analysis set was defined as all participants who completed the study and had safety data available.
Measure: Number; unit: participants
Arm/Group | Alogliptin + Biguanides | Alogliptin + Other
Number analyzed (Participants) | 954 | 109
participants | 26 | 2

2. Primary Outcome: Number of Participants Reporting One or More Serious Adverse Drug Reactions
Description: Serious adverse drug reactions are defined as serious adverse events (SAEs) which are in the investigator's opinion of causal relationship to the study treatment. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The safety analysis was planned to be assessed in alogliptin + biguanides and alogliptin + other arm separately.
Time Frame: Baseline up to 12 months
Population: The safety analysis set was defined as all participants who completed the study and had safety data available.
Measure: Number; unit: participants
Arm/Group | Alogliptin + Biguanides | Alogliptin + Other
Number analyzed (Participants) | 954 | 109
participants | 4 | 0

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at 1 month, 3 months, 6 months, 12 months or final visit (last visit for a participant in the study, up to Month 12) relative to baseline. The efficacy analysis was planned to be assessed in the total alogliptin arm irrespective of biguanide treatment.
Time Frame: Baseline, Months 1, 3, 6, 12, and final assessment (up to Month 12)
Population: The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Groups:
- Alogliptin: Participants who took alogliptin 25 mg, tablets, orally, once daily for up to 12 months as per routine clinical practice were observed.
Arm/Group | Alogliptin
Number analyzed (Participants) | 880
percentage of glycosylated hemoglobin
  Baseline (n = 880) | 7.84 (1.215)
  Change at Month 1 (n = 671) | -0.35 (0.630)
  Change at Month 3 (n = 768) | -0.59 (0.943)
  Change at Month 6 (n = 776) | -0.62 (1.011)
  Change at Month 12 (n = 723) | -0.65 (1.027)
  Change at Final Assessment (n = 880) | -0.58 (1.066)

4. Secondary Outcome: Percentage of Participants of Achieving Objective Glycemic Control
Description: The rate of achieving objective glycemic control in HbA1c level, was calculated at 12 month or final visit (last visit for a participant in the study, up to Month 12). Glycemic control was measured as <8.0%, <7.0%, and <6.0% of glycosylated hemoglobin. The efficacy analysis was planned to be assessed in the total alogliptin arm irrespective of biguanide treatment.
Time Frame: Baseline and final assessment (up to Month 12)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin
Number analyzed (Participants) | 880
percentage of participants
  <8.0% (Baseline) | 62.8
  <8.0% (Final assessment [upto month 12]) | 80.5
  <7.0% (Baseline) | 21.4
  <7.0% (Final assessment [upto month 12]) | 47.2
  <6.0% (Baseline) | 1.4
  <6.0% (Final assessment [upto month 12]) | 5.2

5. Secondary Outcome: Change From Baseline in Fasting Blood Glucose
Description: The change between the fasting blood glucose value collected at 1 month, 3 months, 6 months, 12 months or final visit (last visit for a participant in the study, up to Month 12) relative to baseline. The efficacy analysis was planned to be assessed in the total alogliptin arm irrespective of the biguanide treatment.
Time Frame: Baseline, Months 1, 3, 6, 12, and final assessment (up to Month 12)
Population: The efficacy assessment population was defined as participants who completed the study and had fasting blood glucose data at baseline and post-baseline time points available.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Alogliptin
Number analyzed (Participants) | 253
milligram per deciliter (mg/dL)
  Baseline (n = 253) | 151.8 (48.68)
  Change at Month 1 (n = 160) | -16.7 (40.47)
  Change at Month 3 (n = 198) | -17.1 (47.05)
  Change at Month 6 (n = 189) | -16.0 (44.03)
  Change at Month 12 (n = 186) | -19.1 (40.04)
  Change at final assessment (n = 253) | -17.2 (44.25)

6. Secondary Outcome: Change From Baseline in Fasting Insulin Level
Description: The change between the fasting insulin value collected at 1 month, 3 months, 6 months, 12 months or final visit (last visit for a participant in the study, up to Month 12) relative to baseline. The efficacy analysis was planned to be assessed in the total alogliptin arm irrespective of biguanide treatment.
Time Frame: Baseline, Months 1, 3, 6, 12, and final assessment (up to Month 12)
Population: The efficacy assessment population was defined as participants who completed the study and had fasting insulin data at baseline and post-baseline time points available.
Measure: Mean (Standard Deviation); unit: microunits per milliliter
Arm/Group | Alogliptin
Number analyzed (Participants) | 32
microunits per milliliter
  Baseline (n = 32) | 9.00 (6.712)
  Change at Month 1 (n = 21) | 1.79 (5.485)
  Change at Month 3 (n = 18) | 2.21 (6.305)
  Change at Month 6 (n = 24) | 0.04 (4.913)
  Change at Month 12 (n = 19) | -1.21 (3.711)
  Change at final assessment (n = 32) | -0.25 (5.286)

ADVERSE EVENTS:
Time Frame: Baseline up to 12 months.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Only adverse drug reactions were collected in the safety population.
Arm/Group | Alogliptin + Biguanides | Alogliptin + Other
Serious Adverse Events (participants affected / at risk) | 4/954 | 0/109
Other Adverse Events (participants affected / at risk) | 24/954 | 2/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin + Biguanides (N=954) | Alogliptin + Other (N=109)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin + Biguanides (N=954) | Alogliptin + Other (N=109)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 0
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0
Feeling abnormal (General disorders) | 2 | 0
Weight increased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.